CLINICAL TRIAL: NCT04127604
Title: Post-Hospital Intervention for Veterans With Comorbid Bipolar and Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 19-048; IRB-2019-027 (Other: Providence VA Medical Center)
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder; Substance Use Disorders
Keywords: Bipolar Disorder; Substance Use Disorders; Treatment Adherence; Veterans; Psychosocial intervention
MeSH Terms: conditions — Bipolar Disorder; Substance-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Treatment Adherence Program for Veterans (ITAP-VA) (Experimental): A combination of in-person and phone sessions along with significant other involvement over 6 months post-hospitalization.
  Interventions: Behavioral: Integrated Treatment Adherence Program for Veterans (ITAP-VA)
- Safety Assessment and Follow-up Evaluation (SAFE) (Active Comparator): Enhanced symptom monitoring and safety evaluation over 6 months post-hospitalization.
  Interventions: Behavioral: Safety Assessment and Follow-up Evaluation (SAFE)

INTERVENTIONS:
Behavioral: Integrated Treatment Adherence Program for Veterans (ITAP-VA) — Psychosocial support and treatment to improve treatment adherence, symptoms, and functioning.
  Arms: Integrated Treatment Adherence Program for Veterans (ITAP-VA)
Behavioral: Safety Assessment and Follow-up Evaluation (SAFE) — Measurement-based care assessment and evaluation.
  Arms: Safety Assessment and Follow-up Evaluation (SAFE)

SUMMARY:
This trial aims to evaluate the effectiveness of a novel intervention for Veterans with co-occurring bipolar and substance use disorders following a psychiatric hospitalization. Half of the participants will receive a specialized psychosocial intervention program, while the other half will receive an enhanced safety monitoring program, both provided in addition to their routine care.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the effectiveness of a psychosocial intervention designed to improve treatment adherence in Veterans with comorbid bipolar disorder and substance use disorders (BP-SUD) following a psychiatric hospitalization. Participants will be randomized to either the specialized psychosocial intervention or an enhanced safety monitoring program, both as adjuncts to VA treatment as usual. Veterans with BP-SUD will be recruited from the Providence VAMC inpatient psychiatric unit and assessed at baseline and at 3 (mid-treatment), 6 (post-treatment), and 9-month post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a mood disorder
* Diagnosis of a substance use disorder (drug and/or alcohol)
* Taking at least one psychiatric medication

Exclusion Criteria:

* Unable to speak and read English
* Younger than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Brief Adherence Rating Scale (BARS) | 1 month
  The Brief Adherence Rating Scale (BARS) assesses the percentage of missed medication doses over the past month. The total adherence score ranges from 0% to 100% and higher scores indicate greater adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Metrik, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI; Brandon A Gaudiano, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the studies published, de-identified data will be made available to other qualified researchers on request. The request will be evaluated by the PI and the Co-Investigators to ensure that it meets reasonable standards of scientific integrity.
Supporting Information: Study Protocol, ICF
Time Frame: After all data have been collected and the results of the studies published, de-identified data will be made available to other qualified researchers on request.
Access Criteria: The request will be evaluated by the PI and the Co-Investigators to ensure that it meets reasonable standards of scientific integrity.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT04127604/ICF_000.pdf